CLINICAL TRIAL: NCT00820703
Title: A Randomized, Prospective, Double-blind, Vehicle-controlled, Dose-escalation, Single-center Study of the Safety and Clinical Effect of Nexagon® in the Treatment of Participants With Diabetic Foot Ulcers
Brief Title: The ASCEND Study: A Study to Investigate the Safety and Clinical Effect of Nexagon to Treat Slow Healing Diabetic Foot Ulcers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: For business reasons
Sponsor: OcuNexus Therapeutics, Inc. (Industry)
Responsible Party: Scott Bannan, CoDa Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEX-ULC-003
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Diabetic Foot Ulcer
Keywords: Nexagon; CoDa; ulcer; diabetic; foot
MeSH Terms: conditions — Diabetic Foot; Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Nexagon®
Drug: Nexagon® vehicle

SUMMARY:
Diabetic foot ulcers are sores on the feet that occur in 15% of diabetic patients some time during their lifetime. Once an ulcer develops, the risk of lower-extremity amputation is increased 8-fold in people with diabetes. New treatments that improve the number of ulcers that heal and/or speed up healing are urgently needed. Initial studies with a new drug called Nexagon® (developed by CoDa Therapeutics, Inc.) support the concept that healing of diabetic foot ulcers can be improved with topical application of Nexagon®. Further research will be undertaken to assess the safety and activity of Nexagon® when applied to diabetic foot ulcers at various doses. A proposed randomized controlled trial will randomly allocate (e.g., by the toss of a coin) 24 people with diabetic foot ulcers to Nexagon® (one of three different doses) or vehicle (substance containing no medication) to be applied to their ulcer three times over four weeks. Participants will be followed over four weeks to monitor their response to the treatment, specifically with regards to the amount of healing that occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 and older
2. Female subjects must be a) post-menopausal, b) surgically sterilized, c) practicing abstinence, or d) using hormonal contraceptive, intra-uterine device, diaphragm with spermicide or condom with spermicide for the duration of the study
3. Diabetes mellitus (type I or II) with an HbA1c < 10.0%
4. Diagnosis of neuropathic foot ulcer
5. Cutaneous, full thickness (University of Texas grade A1), below ankle surface ulcer between 0.5 and 5.0 cm2 post-debridement
6. A viable, granulating wound
7. Ulcer present for > 4 weeks prior to study entry
8. An ankle brachial index between 0.70 and 1.3 measured during screening or within three months prior to the Day -14 visit
9. Signed informed consent form

Exclusion Criteria:

1. Decrease or increase in the ulcer size by 30% or more during a14 day "run-in" period
2. Cannot tolerate the off-loading method or comply with standard-of-care
3. An ulcer which shows signs of clinical infection
4. The ulcer to be treated requires operative debridement.
5. An ulcer positive for β-hemolytic streptococcus upon culture.
6. Requirement for total contact casts
7. The ulcer has more than 50% slough, significant necrotic tissue, osteomyelitis, bone, tendon, or capsule exposure
8. Presence of an active systemic or local cancer or tumor of any kind (with the exception of non-melanoma skin cancer)
9. Congestive heart failure NYHA class II - IV
10. Coronary heart disease with STEMI, CABG, or PTCA within the last 6 months
11. Active osteomyelitis of the study foot
12. Active connective tissue disease
13. Acute Charcot's neuroarthropathy as determined by clinical and/or radiographic examination
14. Treatment with systemic corticosteroids (
15. Previous or current radiation therapy to the distal lower extremity or likelihood to receive this therapy during study participation
16. Pregnancy or lactation
17. eGFR < 25 mL/min
18. Poor nutritional status defined as an albumin < 25 g/L
19. Significant peripheral edema
20. Known prior inability to complete required study visits during study participation
21. A psychiatric condition (e.g., suicidal ideation) or chronic alcohol or drug abuse problem, determined from the subject's medical history, which, in the opinion of the Investigator, may pose a threat to subject compliance
22. Use of a platelet-derived growth factor within the 28 days prior to screening
23. Use of any investigational drug or therapy within the 28 days prior to screening
24. Any other factor which may, in the opinion of the Investigator, compromise participation and follow-up in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and clinical effect of Nexagon® administered topically to diabetic foot ulcers.

SECONDARY OUTCOMES:
To select the optimal dose(s) which can be used in future trials of Nexagon® in diabetic foot ulcers
To pilot the collection of data that may be considered useful in planning future studies of Nexagon® administered topically to diabetic foot ulcers.

CONTACTS AND LOCATIONS:
Locations (1):
- Middlemore Hospital, Auckland, Auckland, New Zealand